CLINICAL TRIAL: NCT00070382
Title: A Randomized, Open-Label, Multicenter Study Of Darbepoetin Alfa Administered Once Every Two Weeks (Q2W) Compared With rHuEPO Administered Once Every Week (QW) For The Treatment Of Anemia In Subjects With Non-Myeloid Malignancies Receiving Multiple Chemotherapy
Brief Title: Darbepoetin Alfa Compared With Epoetin Alfa in Treating Anemia in Patients Receiving Chemotherapy for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000333213; UCLA-0306021; AMGEN-20030125
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-08

CONDITIONS: Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorder; Multiple Myeloma and Plasma Cell Neoplasm; Precancerous/Nonmalignant Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: anemia; unspecified adult solid tumor, protocol specific; Waldenstrom macroglobulinemia; monoclonal gammopathy of undetermined significance; extramedullary plasmacytoma; isolated plasmacytoma of bone; refractory multiple myeloma; primary systemic amyloidosis; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; post-transplant lymphoproliferative disorder; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; recurrent adult T-cell leukemia/lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; recurrent adult Hodgkin lymphoma; stage I adult Hodgkin lymphoma; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; T-cell large granular lymphocyte leukemia; refractory chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; prolymphocytic leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; recurrent mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma
MeSH Terms: conditions — Anemia; Leukemia; Lymphoma; Lymphoproliferative Disorders; Multiple Myeloma; Neoplasms, Plasma Cell; Precancerous Conditions; Waldenstrom Macroglobulinemia; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, T-Cell, Cutaneous; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Mycosis Fungoides; Sezary Syndrome; Hodgkin Disease; Leukemia, Large Granular Lymphocytic; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Mantle-Cell | interventions — Darbepoetin alfa; Epoetin Alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Darbepoetin alfa (Experimental): darbepoetin alfa administered once every two weeks at a dose of 200 ug over a 16 week treatment period.
  Interventions: Drug: darbepoetin alfa
- Epoetin alfa (Active Comparator): epoetin alfa administered at 40,000 unites, once per week over a 16-week treatment period.
  Interventions: Drug: epoetin alfa

INTERVENTIONS:
Drug: darbepoetin alfa — darbepoetin alfa administered at a dose of 200ug once every 2 weeks over a 16-week treatment period
  Arms: Darbepoetin alfa
Drug: epoetin alfa — epoetin alfa administered at a dose of 40,000U once every week over a 16-week treatment period
  Arms: Epoetin alfa

SUMMARY:
RATIONALE: Darbepoetin alfa and epoetin alfa may stimulate red blood cell production and treat anemia in patients who are receiving chemotherapy. It is not yet known whether darbepoetin alfa is more effective than epoetin alfa in treating patients with anemia.

PURPOSE: Randomized phase III trial to compare the effectiveness of darbepoetin alfa with that of epoetin alfa in treating anemia in patients who are receiving chemotherapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the efficacy of darbepoetin alfa vs epoetin alfa for anemia in patients with non-myeloid malignancies receiving chemotherapy.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to screening hemoglobin concentration (less than 10.0 g/dL vs 10.0-11.0 g/dL) and type of concurrent chemotherapy (platinum-based vs non-platinum-based). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive darbepoetin alfa subcutaneously (SC) every other week for 12 weeks (i.e., on weeks 1, 3, 5, 7, 9, and 11).
* Arm II: Patients receive epoetin alfa SC once weekly for 12 weeks. Patients are followed at 1 and 3 weeks .

PROJECTED ACCRUAL: A total of 600 patients (300 per treatment arm) will be accrued for this study within 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a non-myeloid malignancy
* Currently receiving or planning to receive at least 8 weeks of cyclic cytotoxic chemotherapy
* Hemoglobin no greater than 11.0 g/dL
* 18 and over
* ECOG 0-2
* Bilirubin less than 2 times upper limit of normal (ULN)
* Creatinine less than 2 times ULN
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* More than 30 days since prior darbepoetin alfa or epoetin alfa
* More than 30 days since prior participation in investigational device or drug trials

Exclusion Criteria:

* The following diagnoses are excluded:

  * Acute myeloid leukemia
  * Chronic myeloid leukemia
  * Acute lymphoblastic leukemia
  * Hairy cell leukemia
  * Burkitt's lymphoma
  * Lymphoblastic lymphoma
* other primary hematologic disorder that would cause anemia (e.g., sickle cell anemia)
* angina
* congestive heart failure
* New York Heart Association class III or IV heart disease
* hypertension
* cardiac arrhythmia
* other unstable or uncontrolled disease or condition that would affect cardiac function
* pregnant or nursing
* known seizure disorder
* known sensitivity to study agents
* clinically significant inflammatory disease (e.g., rheumatoid arthritis or Crohn's disease)
* confirmed neutralizing antibodies to epoetin alfa
* other disorder that would preclude study compliance or giving informed consent
* other concurrent epoetin alfas
* prior randomization to this study
* other concurrent investigational agents or procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2003-08; Primary Completion 2003-11 (Actual)

PRIMARY OUTCOMES:
Compare Efficacy of darbepoetin alfa with Epoetin Alfa as measured by the incidence of red blood cell transfusions. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John A. Glaspy, MD, MPH, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California, United States

REFERENCES:
- [Result] 20030125 Study Group Trial; Glaspy J, Vadhan-Raj S, Patel R, Bosserman L, Hu E, Lloyd RE, Boccia RV, Tomita D, Rossi G. Randomized comparison of every-2-week darbepoetin alfa and weekly epoetin alfa for the treatment of chemotherapy-induced anemia: the 20030125 Study Group Trial. J Clin Oncol. 2006 May 20;24(15):2290-7. doi: 10.1200/JCO.2005.03.8570. PMID 16710026